CLINICAL TRIAL: NCT05328440
Title: Treatment of Dalpiciclib Combined With Pyrotinib for Trastuzumab-sensitive HER2+ Advanced Breast Cancer: a Single Arm, Dual Cohort, Prospective, Open Phase II Exploratory Study
Brief Title: Treatment of Dalpiciclib Combined With Pyrotinib for Trastuzumab-sensitive HER2+ Advanced Breast Cancer(DAP-Her-02)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Min Yan, MD, Chief Physician, Henan Cancer Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-BC-II-037
Record Dates: First submitted 2022-03-14; First posted 2022-04-14 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Breast Neoplasms
Keywords: HER2-positive MBC
MeSH Terms: conditions — Breast Neoplasms | interventions — pyrotinib; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): HR-positive/HER2-positive MBC
  Interventions: Drug: Pyrotinib Maleate; Drug: Dalpiciclib Isethionate Tablets; Drug: Fulvestrant
- Arm B (Experimental): HR-negative/HER2-positive MBC
  Interventions: Drug: Pyrotinib Maleate; Drug: Dalpiciclib Isethionate Tablets; Drug: Inetetamab

INTERVENTIONS:
Drug: Pyrotinib Maleate — once a day, 125mg each time, taking for 3 weeks, stopping for 1 week, 4 weeks as a cycle. It is recommended to take medicine at about the same time every day, take it with warm water, and fast at least 1 hour before and after taking medicine
  Other Names: Pyrotinib
Drug: Dalpiciclib Isethionate Tablets — 400mg once a day, oral administration within 30 minutes after breakfast, continuous administration for 28 days as a cycle
  Other Names: SHR6390
Drug: Inetetamab — the initial dose is 8mg / kg and the subsequent dose is 6mg / kg. It is administered intravenously for 21 days.
  Arms: Arm B
Drug: Fulvestrant — fluvestrant is administered intravenously on the 1/15 day of the first cycle, and then on the first day of each cycle, 500mg / time, intravenously
  Arms: Arm A

SUMMARY:
Based on different HR status, we explored the efficacy and safety of Pyrotinib and Dalpiciclib Isethionate Tablets based combination regimen in the first-line treatment of HER2 + MBC.

DETAILED DESCRIPTION:
Cyclin D-CDK4/6-RB-E2F signaling pathway regulates the transformation of breast cancer cells from stage G1 to S, and plays an important role in the proliferation of breast cancer cells. HER2 protein regulates proliferation of breast cancer cells through PI3K/AKT signaling pathway. HER2 positive breast cancer patients need anti HER2 therapy. Data indicate that HER2 positive breast cancer patients often express cyclin D1 and E1, suggesting that anti HER2 therapy can synergy with CDK4/6 inhibitors.

A preclinical study shows that the combination of CDK4/6 inhibitor Dulcie and anti HER2 drug pyrrolidone can effectively reduce the phosphorylation of AKT and HER3, thereby promoting the apoptosis of HER2 positive breast cancer cells and achieving the purpose of inhibiting tumor.

In the clinical study of na-phere 2, piperacillin combined with trastuzumab, patuzumab and fluvestrant can significantly inhibit the expression of Ki67. MonarcHER study shows that the treatment of patients with advanced HR+HER2+ breast cancer after the failure of anti HER2+ is better than conventional chemotherapy plus anti HER2 therapy. The successful challenge of traditional chemotherapy is the opening of a new chapter in the treatment of HR+/HER2+. In 2021, ESMO 276P reported the interim data of darcilil combined with pyrroltinib in the first-line / second-line treatment of MBC. HR -, HER2 + MBC ORR can reach 81.8%, and the safety is controllable.

Based on different HR status, we explored the efficacy and safety of Pyrotinib and Dalpiciclib Isethionate Tablets based combination regimen in the first-line treatment of HER2 + MBC.

ELIGIBILITY:
Inclusion Criteria:

1. Premenopausal / perimenopausal / postmenopausal women who aged ≥ 18 years
2. Suffering from non resectable locally advanced recurrent breast cancer or metastatic breast cancer
3. group A: Women who have breast cancer histopathologically confirmed by positive estrogen receptor (ER; >10%), positive progesterone receptor (PR; >1%), and positive human epidermal growth factor receptor 2 (HER2) according to the 2018 American Society of Clinical Oncology/College of American Pathologists (ASCO/CAP) human epidermal growth factor receptor 2 (HER2) guideline. The pathological laboratory confirmed that the immunohistochemical (IHC) score was 3 +, or 2 +, and the in situ hybridization (ISH) test was positive (ISH amplification rate ≥ 2.0); (New) the end of trastuzumab treatment in the adjuvant treatment stage > 12 months, recurrence and metastasis, or no trastuzumab treatment in the early stage; No adjuvant endocrine therapy or postoperative adjuvant endocrine therapy > 24 months; Premenopausal or perimenopausal patients need to be combined with ofs (OFS includes bilateral ovariectomy or GnRHa drugs); group B: Women who have breast cancer histopathologically confirmed by negative estrogen receptor (ER), negative progesterone receptor (PR; <1%), and positive human epidermal growth factor receptor 2 (HER2) according to the 2018 American Society of Clinical Oncology/College of American Pathologists (ASCO/CAP) human epidermal growth factor receptor 2 (HER2) guideline. The pathological laboratory confirmed that the immunohistochemical (IHC) score was 3 +, or 2 +, and the in situ hybridization (ISH) test was positive (ISH amplification rate ≥ 2.0); (New) the end of trastuzumab treatment in the adjuvant treatment stage > 12 months, recurrence and metastasis, or no trastuzumab treatment in the early stage;
4. No previous systematic treatment for advanced diseases
5. at least one measurable lesion or only bone metastasis according to RECIST 1.1.
6. Eastern Cooperative Oncology Group (ECOG) performance status 0～1.
7. The patient must be able to swallow oral drugs
8. The functional level of organs must meet the following requirements:

   a) Bone marrow function i) Absolute neutrophil count（ANC）≥1.5×109/L (no use of growth factor within 14 days) ii) Platelet count（PLT）≥100×109/L (no corrective treatment within 7 days) iii) Hemoglobin level（Hb）≥100 g/L (no corrective treatment within 7 days) b) Liver and kidney function i) Total bilirubin（TBIL）≤1.5 upper limit of normal value (ULN) ii) Alanine transaminase (ALT) and aspartate transaminase (AST) ≤3×ULN iii) Blood urea nitrogen (BUN) and creatinine ≤1.5×ULN and creatinine clearance≥50 mL/min (Cockcroft-Gault formula); c) Color Doppler echocardiography: Left ventricular ejection fraction ≥50% d) 12-lead electrocardiography: QTc interval ≤480 ms
9. Volunteers to participate in the study, provision of signed informed consent, good compliance and willingness to cooperate with follow-ups.

Exclusion Criteria:

1. Patients with symptomatic brain metastasis;
2. Unable to swallow, chronic diarrhea and intestinal obstruction, there are many factors affecting drug use and absorption;
3. patient who received radiotherapy, chemotherapy, surgery (excluding local puncture) or molecular targeted therapy within 4 weeks before admission; those who received anti-tumor endocrine therapy after screening period;
4. Participated in other drug clinical trials within 4 weeks before admission;
5. Tyrosine kinase inhibitors targeting HER2 (Neratinib, Lapatinib, pyrotinib, etc.) have been used or are being used in the past;
6. Patients previously treated with any CDK4 / 6 inhibitor;
7. Those who have other malignant tumors (with the exception of healed cervical carcinoma in situ) occurring in the past 5 years;
8. Those who are known to have a history of allergy to the component of study drugs; those who have a history of immunodeficiency, including positive detection of human immunodeficiency virus, hepatitis C virus, active hepatitis B or other acquired, congenital immunodeficiency diseases, or organ transplantation;
9. Those who had suffered from any heart disease, including arrhythmia which requires drug treatment or is of clinical significance; myocardial infarction; heart failure; and any other heart disease judged by the investigator as unsuitable for this trial;
10. Pregnant and lactating women; fertile women who provide positive results of baseline pregnancy test; women of childbearing age who are unwilling to take effective contraceptive measures during the whole study period;
11. If the accompanying diseases (including, but not limited to, severe hypertension, severe diabetes, and active infection, which cannot be controlled by drugs) that would be a potential hazard to participant's health, or affect the completion of the study as per investigator's judgement;
12. Moderate infection occurs within 4 weeks before the first administration (e.g. intravenous drip of antibiotics, antifungal or antiviral drugs according to clinical criteria), fever（> 38.5 ℃） of unknown origin occurs during the screening period/before the first administration.
13. A clear history of neurological or psychiatric disorders, including epilepsy or dementia.
14. Researchers believe that patients are not suitable for any other situation in this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-05-20 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
PFS (Progression-Free survival) | up to 2 years
  From the date into this study (signed ICF) to tumor progression or death.

SECONDARY OUTCOMES:
ORR (Objective control rate) | up to 2 years
  The rate of CR and PR, determined using RECIST v1.1 criteria
Overall survival (OS) | up to 2 years
  It refers to the length of time from the start of treatment to the death of the patient

OTHER OUTCOMES:
Subject safety | Through study completion,an average of 4 year
  Number of Adverse Events using NCI CTCAE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Min Yan, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identificationare available following article publication.
Supporting Information: Study Protocol
Time Frame: five years after publication
Access Criteria: Please contact Central contact person by Email